CLINICAL TRIAL: NCT06211608
Title: Ultrasound Assessment of Uterine and Endometrium Volume in Women With PCOS and HPOD
Brief Title: Uterine and Endometrial Volume in PCOS and HPOD
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, PhD, MD, Jagiellonian University
Other Study IDs: 118.6120.53.2023
Record Dates: First submitted 2024-01-07; First posted 2024-01-18 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Anovulation; Irregular Menses
Keywords: Uterine morphology; PCOS; Hypothalamic-pituitary-ovarian axis dysfunction; Endometrial volume
MeSH Terms: conditions — Anovulation; Menstruation Disturbances

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Polycystic ovary syndrome (PCOS)
  Interventions: Diagnostic Test: Two-dimensional and three-dimensional ultrasound of the female reproductive organ
- Arm 2: Hypothalamic-pituitary-ovarian axis dysfunction (HPOD)
  Interventions: Diagnostic Test: Two-dimensional and three-dimensional ultrasound of the female reproductive organ

INTERVENTIONS:
Diagnostic Test: Two-dimensional and three-dimensional ultrasound of the female reproductive organ — Two-dimensional and three-dimensional ultrasound of the female reproductive organ using a Samsung WS80A or Samsung HERA W10 ultrasound device with a transvaginal or transabdominal transducer

SUMMARY:
Group II causes of anovulation according to the World Health Organization include polycystic ovary syndrome (PCOS) and the less common dysfunction of the hypothalamic-pituitary-ovarian axis (HPOD). Assessment of ovarian volume, number and morphology of ovarian follicles is essential in the diagnosis of menstrual disorders, including PCOS and HPOD. However, the uterus is a target organ for steroid hormones, and the assessment of uterine size and endometrial morphology may also be of clinical importance. While ultrasonographic features of the ovaries in PCOS have been described and constitute one of the diagnostic criteria for the syndrome (Rotterdam criteria), there is little data on uterine volume in women with PCOS and HPOD. The aim is to compare ultrasound i) uterine volume and ii) endometrial volume among women with PCOS and women with HPOD.

DETAILED DESCRIPTION:
Group II causes of anovulation according to the World Health Organization include polycystic ovary syndrome (PCOS) and the less common dysfunction of the hypothalamic-pituitary-ovarian axis (HPOD). The exact etiology of both entities is unknown. The diagnosis of PCOS requires meeting the Rotterdam criteria. HPOD, in turn, is considered a functional disorder of the axis, related to lifestyle factors, and the diagnosis is made after excluding identifiable causes of ovulation disorders. Assessment of ovarian volume, number and morphology of ovarian follicles is essential in the diagnosis of menstrual disorders, including PCOS and HPOD. However, the uterus is a target organ for steroid hormones, and the assessment of uterine size and endometrial morphology may also be of clinical importance. The dimensions and volume of the uterus and endometrium may influence the clinical pregnancy rate in women undergoing assisted reproductive technologies. Both too small and too large sizes and volumes of the uterus may reduce the rate of clinical pregnancies. Too small dimensions may result from hypoestrogenism, while excessive size may be the result of estrogen-progesterone imbalance accompanying PCOS, increased uterine vascularity, as well as estrogen-dependent changes in the uterine myometrium, such as adenomyosis. Similarly, too "thin" endometrium and too thick (cystic) endometrium may reduce the receptivity of the endometrium. While ultrasonographic features of the ovaries in PCOS have been described and constitute one of the diagnostic criteria for the syndrome (Rotterdam criteria), there is little data on uterine volume in women with PCOS and HPOD. The aim is to compare ultrasound uterine volume and endometrial volume among women with PCOS and women with HPOD. The volume of the uterus will be determined according to the formula: V = (π/6) × length × width × height (in cm and given in ml). The volume of the endometrium will also be measured according to a similar formula.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 years
* no previous diagnosis and treatment due to menstrual disorders or infertility

Exclusion Criteria:

* previous ovarian surgery
* use of drugs that disturb the functions of the hypothalamic-pituitary-ovarian axis
* uterine tumors

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include women diagnosed in the Clinical Department of Gynecological Endocrinology and Gynecology of the University Hospital inn Krakow, Poland, and the Gynecological Endocrinology Clinic due to menstrual disorders or infertility due to ovulation disorders. The size of the group is estimated at 300 women aged 18-45.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Uterine volume | 12 months
  Comparison of uterine volume in ml calculated using the presented formula in both arms of the study
Endometrium volume | 12 months
  Comparison of endometrial volume in ml calculated using the presented formula in both arms of the study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jach, Prof., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No